CLINICAL TRIAL: NCT02289807
Title: Prospective Non-inferior Clinical Trial Comparing Concurrent Chemoradiotherapy or Radiotherapy Alone in Patients With Intermediate Risk Nasopharyngeal Carcinoma in Intensity-modulated Radiotherapy Era
Brief Title: Concurrent Chemotherapy in Intermediate Risk Patients Treated With Intensity-modulated Radiotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSYCC-2014-11
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2014-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Concurrent chemoradiotherapy; intermediate risk; intensity-modulated radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RT group (Experimental): intensity modulated-radiotherapy (IMRT) alone Patients receive intensity modulated-radiotherapy (IMRT) alone
  Interventions: Radiation: IMRT
- CCRT group (Active Comparator): IMRT and concurrent cisplatin Patients receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles
  Interventions: Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Cisplatin — concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles during IMRT
  Arms: CCRT group
Radiation: IMRT — Intensity modulated-radiotherapy (IMRT) is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor

SUMMARY:
Currently, concurrent chemoradiotherapy with/without sequential chemotherapy is the standard treatment modality for intermediate risk NPC (stage II and T3N0M0) according to the National Comprehensive Cancer Network guideline. However these recommendations were based on the evidence in the two-dimensional conventional radiotherapy (2DCRT) era. The introduction of intensity-modulated radiotherapy (IMRT) in NPC treatment has brought substantial better treatment outcomes than 2DCRT. It has been questioned whether additional concurrent chemotherapy is still necessary for intermediate risk NPC within the excellent framework of IMRT. hus, we jointly conduct the first non-inferior randomized trial to determine the value of concurrent chemotherapy with cisplatin for intermediate risk NPC patients treated with IMRT. Given the results of clinical studies mentioned above, we decide to adopt the concurrent regimen to be cisplatin 100 mg/m2 on day 1, 22, 43

DETAILED DESCRIPTION:
Patients Patients with non-keratinizing NPC T1-2N1M0/T2-3N0M0 (UICC/AJCC 7th edition) are randomly assigned to receive CCRT or RT alone. Patients in CCRT group receive cisplatin 100 mg/m² every 3 weeks for 3 cycles, concurrently with intensity-modulated radiotherapy (IMRT). IMRT is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor. Our primary endpoint is failure-free survival(FFS). Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), distant failure-free survival (D-FFS) rates and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).

Tumor staged as T1-2N1/T2-3N0(according to the 7th AJCC edition). No evidence of distant metastasis (M0). Satisfactory performance status: Karnofsky scale (KPS) ≥ 70. Adequate marrow: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.

Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN.

Adequate renal function: creatinine clearance ≥ 60 ml/min. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

Neck lymph node with extracapsular spread. Maximal axial diameter of neck lymph node ≥30mm, positive neck lymph node at level IV and/or Vb.

Pretherapy plasma EBV DNA level ≥4000 copy/ml. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.

Age > 70 or < 18. Treatment with palliative intent. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.

Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).

History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).

Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2020-08 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3 Year
  Failure-free survival rate is calculated from the date of randomization to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3 Year
  Overall survival is calculated from randomization to death from any cause
Locoregional failure-free survival | 3 Year
  Locoregional failure-free survival is calculated from randomization to the first locoregional failure.
Distant failure-free survival | 3 Year
  Distant failure-free survival is calculated from randomization to the first remote failure.
Number of participants with adverse events | 3 Year
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chua DT, Sham JS, Kwong DL, Au GK. Treatment outcome after radiotherapy alone for patients with Stage I-II nasopharyngeal carcinoma. Cancer. 2003 Jul 1;98(1):74-80. doi: 10.1002/cncr.11485. PMID 12833458
- [Background] Xiao WW, Han F, Lu TX, Chen CY, Huang Y, Zhao C. Treatment outcomes after radiotherapy alone for patients with early-stage nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2009 Jul 15;74(4):1070-6. doi: 10.1016/j.ijrobp.2008.09.008. Epub 2009 Feb 21. PMID 19231110
- [Background] Chen QY, Wen YF, Guo L, Liu H, Huang PY, Mo HY, Li NW, Xiang YQ, Luo DH, Qiu F, Sun R, Deng MQ, Chen MY, Hua YJ, Guo X, Cao KJ, Hong MH, Qian CN, Mai HQ. Concurrent chemoradiotherapy vs radiotherapy alone in stage II nasopharyngeal carcinoma: phase III randomized trial. J Natl Cancer Inst. 2011 Dec 7;103(23):1761-70. doi: 10.1093/jnci/djr432. Epub 2011 Nov 4. PMID 22056739
- [Background] Song CH, Wu HG, Heo DS, Kim KH, Sung MW, Park CI. Treatment outcomes for radiotherapy alone are comparable with neoadjuvant chemotherapy followed by radiotherapy in early-stage nasopharyngeal carcinoma. Laryngoscope. 2008 Apr;118(4):663-70. doi: 10.1097/MLG.0b013e3181626cfe. PMID 18216741
- [Background] Chua DT, Ma J, Sham JS, Mai HQ, Choy DT, Hong MH, Lu TX, Au GK, Min HQ. Improvement of survival after addition of induction chemotherapy to radiotherapy in patients with early-stage nasopharyngeal carcinoma: Subgroup analysis of two Phase III trials. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1300-6. doi: 10.1016/j.ijrobp.2006.02.016. Epub 2006 Jun 5. PMID 16750333
- [Background] Xu T, Hu C, Wang X, Shen C. Role of chemoradiotherapy in intermediate prognosis nasopharyngeal carcinoma. Oral Oncol. 2011 May;47(5):408-13. doi: 10.1016/j.oraloncology.2011.03.008. Epub 2011 Apr 2. PMID 21459659
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Peng G, Wang T, Yang KY, Zhang S, Zhang T, Li Q, Han J, Wu G. A prospective, randomized study comparing outcomes and toxicities of intensity-modulated radiotherapy vs. conventional two-dimensional radiotherapy for the treatment of nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):286-93. doi: 10.1016/j.radonc.2012.08.013. Epub 2012 Sep 17. PMID 22995588
- [Background] Lee AW, Ng WT, Chan LL, Hung WM, Chan CC, Sze HC, Chan OS, Chang AT, Yeung RM. Evolution of treatment for nasopharyngeal cancer--success and setback in the intensity-modulated radiotherapy era. Radiother Oncol. 2014 Mar;110(3):377-84. doi: 10.1016/j.radonc.2014.02.003. Epub 2014 Mar 11. PMID 24630534
- [Background] Su SF, Han F, Zhao C, Chen CY, Xiao WW, Li JX, Lu TX. Long-term outcomes of early-stage nasopharyngeal carcinoma patients treated with intensity-modulated radiotherapy alone. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):327-33. doi: 10.1016/j.ijrobp.2010.09.011. Epub 2010 Oct 29. PMID 21035959
- [Background] Tham IW, Lin S, Pan J, Han L, Lu JJ, Wee J. Intensity-modulated radiation therapy without concurrent chemotherapy for stage IIb nasopharyngeal cancer. Am J Clin Oncol. 2010 Jun;33(3):294-9. doi: 10.1097/COC.0b013e3181d2edab. PMID 20395788
- [Background] Luo S, Zhao L, Wang J, Xu M, Li J, Zhou B, Xiao F, Long X, Shi M. Clinical outcomes for early-stage nasopharyngeal carcinoma with predominantly WHO II histology treated by intensity-modulated radiation therapy with or without chemotherapy in nonendemic region of China. Head Neck. 2014 Jun;36(6):841-7. doi: 10.1002/hed.23386. Epub 2013 Oct 4. PMID 23720240